CLINICAL TRIAL: NCT04257396
Title: Multicentre Randomized Controlled Trial Of A Carbon-Fibre Adjustable Reusable Accessory (CARA) For Supine Breast Positioning To Reduce Toxicity In Whole Breast Adjuvant Radiotherapy
Brief Title: Carbon-Fibre Accessory (CARA) for Supine Breast Positioning to Reduce Toxicity in Whole Breast Radiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Cheryl Duzenli, Medical Physicist, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: H19-03343
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Adjuvant Radiotherapy for Breast Cancer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Skin assessments carried out by blinded observers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 CARA Positioning (Experimental): Arm 1 patients will receive CARA breast support. The known benefits to using CARA for breast positioning are reduction in IMF skin folds during treatment, reduction in breast separation, and reduction in V50% body, V105% body and lung V20 Gy in treatment planning. No known risks to using CARA have been identified.
  Interventions: Device: Carbon-Fibre Adjustable Reuseable Accessory (CARA)
- Arm 2 Standard of Care (No Intervention): Arm 2 patients will not receive CARA breast support. Patients in arm 2 may be treated with no breast support, a small foam wedge, a thermoplastic shell or alternate supine breast support method according to the current standard of care at the treating centre. These methods have entered RT clinical practice over decades of practice without published evidence of impact on rates of MD. Published rates of MD for the control arm thus pertain to a cross section of these methods. The control arm of this study will look at all of these methods combined. There may be centre specific preference for the control method and stratification by centre will be done.

INTERVENTIONS:
Device: Carbon-Fibre Adjustable Reuseable Accessory (CARA) — Breast support device having a carbon-fibre breast cradle for supine patient positioning.
  Arms: Arm 1 CARA Positioning

SUMMARY:
This trial is designed to assess the efficacy of a novel carbon-fibre adjustable reusable accessory (CARA) for breast support to reduce skin toxicity and unwanted normal tissue dose in comparison to the current clinical standard for supine breast support during whole breast RT.

DETAILED DESCRIPTION:
This study is designed to assess the effectiveness of utilizing the CARA positioning device for reducing the incidence and severity of acute skin reactions in the infra-mammary fold in patients undergoing WBRT. Secondary outcomes include patient reported outcomes and dose to normal body tissue and organs at risk. This is a randomized controlled trial. Participants will be randomly assigned to the following two arms:

Arm 1 patients will receive CARA breast support. The known benefits to using CARA for breast positioning are reduction in IMF skin folds during treatment, reduction in breast separation, and reduction in V50% body, V105% body and lung V20 Gy in treatment planning. No known risks to using CARA have been identified.

Arm 2 patients will not receive CARA breast support. Patients in arm 2 may be treated with no breast support, a small foam wedge, a thermoplastic shell or alternate supine breast support method according to the current standard of care at the treating centre. These methods have entered RT clinical practice over decades of practice without published evidence of impact on rates of MD. Published rates of MD for the control arm thus pertain to a cross section of these methods. The control arm of this study will look at all of these methods combined. There may be centre specific preference for the control method and stratification by centre will be done.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older.
* Able to provide informed consent
* ECOG performance status 0 - 2
* Stage 0-3 invasive breast cancer or DCIS scheduled to received adjuvant radiotherapy to the whole breast
* Any infra-mammary skin fold of >= 0.5 cm in the supine treatment position and/or palpable lateral breast tissue falling posterior to the mid-axilla line while in supine or treatment position.

Exclusion Criteria:

* Inability to give informed consent or comply with experimental arm of trial
* Previous RT to either breast or to the chest
* Planned boost to infra mammary area
* Use of Mepitel while on treatment
* Failure to heal surgical wound or significant post-operative wound infection
* Presence of significant connective tissue disease (e.g. systemic sclerosis, SLE)
* Known radiation hypersensitivity phenotype (e.g. ataxia telangiectasia etc.)
* Breast reconstruction
* Planned partial breast irradiation, unless the treated area includes the infra-mammary fold

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rates of moist desquamation in the infra-mammary fold | up to two weeks post radiotherapy
  Presence or absence of moist desquamation

SECONDARY OUTCOMES:
Severity of moist desquamation (MD) in the IMF | up to two weeks post radiotherapy
  Scoring of patch versus confluent moist desquamation
NCI CTAE V 4 skin toxicity | up to two weeks post radiotherapy
  overall breast skin reaction scores
Ipsilateral Lung V20 Gy | prior to first treatment, 1 week
  Planned volume of ipsilateral lung receiving >=20 Gy
Heart V25Gy | prior to first treatment, 1 week
  Planned volume of heart receiving 25Gy for left breast patients
V50% body and V105% body | prior to first treatment, 1 week
  planned volume of body receiving >=50% and >=105% of the prescribed dose
Dose-area predictor of moist desquamation | through study completion, up to 5 weeks
  Measured dose to skin using radio-chromic film on three treatment fractions
Workflow | through study completion, up to 5 weeks
  Measured time for treatment setup
Reproducibility of treatment setup | through study completion, up to 5 weeks
  Shifts in patient position measured with daily and weekly imaging
Patient Reported Skin Toxicity | through study completion, up to 7 weeks
  Questionnaire with 11 questions for patients to report pain, fatigue, skin reaction, open skin, sleep and work interruption, and comfort during treatment on 4 point scale
User experience with the setup technique | through study completion, up to 5 weeks
  Survey with 5 questions using a 4 point scale to collect radiation therapist assessment of ease of use and overall satisfaction with the setup method

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - BC Cancer, Prince George, British Columbia
  - BC Cancer, Surrey, British Columbia
  - BC Cancer, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malhotra A, Chan EK, Nichol A, Duzenli C. Spatial dose-distribution-based risk mapping to predict moist desquamation in breast radiotherapy. Phys Med Biol. 2025 May 27;70(11). doi: 10.1088/1361-6560/add985. PMID 40373801
- [Derived] Duzenli C, Chan EK, Bergman AM, Grahame S, Singer J, Burns L, Olson RA. A novel carbon-fibre adjustable reusable accessory (CARA) for supine breast positioning to reduce toxicity in breast adjuvant radiotherapy: a study protocol for a multicentre phase III randomized controlled trial. BMC Cancer. 2022 Jun 20;22(1):673. doi: 10.1186/s12885-022-09759-y. PMID 35725457